CLINICAL TRIAL: NCT00489086
Title: A Phase II Single Arm Open-Label Clinical Trial of Chemotherapy of BCC's With Tazarotene 0.1% in Subjects With Basal Cell Nevus Syndrome
Brief Title: Topical Tazarotene in Treating Patients With Basal Cell Skin Cancer and Basal Cell Nevus Syndrome on the Face
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000551655; R01CA109584 (NIH); NCT00500643 (obsolete NCT alias)
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Neoplastic Syndrome
Keywords: nevoid basal cell carcinoma syndrome; basal cell carcinoma of the skin
MeSH Terms: conditions — Neoplasms; Basal Cell Nevus Syndrome; Carcinoma, Basal Cell | interventions — tazarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tazarotene Cream (Other): Open label
  Interventions: Drug: tazarotene

INTERVENTIONS:
Drug: tazarotene — Tazarotene is a member of the acetylenic class of retinoids.
  Other Names: tazorac

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as tazarotene, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying topical tazarotene to see how well it works in treating patients with basal cell skin cancer and basal cell nevus syndrome on the face.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether topical tazarotene, administered over a period of 18 months as a chemopreventive agent, reduces the incidence of basal cell carcinomas (BCCs) on treated skin in patients with basal cell nevus syndrome (BCNS).
* Expand and refine chemopreventive strategies in patients with BCNS who are at high risk for the development of BCCs.

OUTLINE: This is an open-label, multicenter study.

Patients apply topical tazarotene cream to the face once daily for 18 months in the absence of unacceptable toxicity.

ELIGIBILITY:
List of Inclusion Criteria:

1. Study subjects must have at least one basal cell carcinoma ≥ 3mm in diameter (target lesion) on any area of the skin except the face, chest, and back (and not impinging on vital sites) diagnosed clinically by a Study Investigator at the baseline visit.
2. Study subjects must meet diagnostic criteria for basal cell nevus syndrome including major criterion #1 plus one additional major criterion or two of the minor criteria outlined in Table I. A first degree relative would satisfy BCNS diagnostic criteria with any two major criteria or any single major plus two minor criteria.

Table I. BCNS Diagnostic Criteria

Major criteria

1. More than 2 BCCs or one under the age of 20 years
2. Odontogenic keratocysts of the jaw proven by histology
3. Three or more palmar and/or plantar pits
4. Bilamellar calcification of the falx cerebri (if less than 20 years old)
5. Fused, bifid, or markedly splayed ribs.
6. First degree relative with basal cell nevus syndrome (BCNS)
7. PTCH1 gene mutation in normal tissue*

Minor criteria

1. Macrocephaly determined after adjustment for height
2. Congenital malformations: cleft lip or palate, frontal bossing, "coarse face."
3. Skeletal abnormalities: Sprengel deformity, marked pectus deformity
4. Radiological abnormalities: bridging of the sella turcica, vertebral anomalies such as hemivertebrae, fusion or elongation of the vertebral bodies.
5. Ovarian fibroma
6. Medulloblastoma

3.The subject is from 18-75 years of age, inclusive.

4. If the subject is female and of child-bearing potential (women are considered not of childbearing potential if they are at least 2 years post-menopausal and/or surgically sterile), she:

i. has been using adequate contraception (abstinence, IUD, birth control pills, or spermicidal gel with diaphragm or condom) since her last menses and will use adequate contraception during the study, and ii. is not lactating, and iii. has documented one negative serum pregnancy test within 14 days prior to study entry.

5. The subject is willing to abstain from application of non-study topical medications to the skin of the face for the duration of the study, including prescription and over the counter preparations.

6. The subject is willing not to have targeted BCCs treated by their PSCP unless the BCCs are documented by Study Investigators, preferably on two separate visits, except when the PSCP believes that delay in treatment potentially might compromise the health of the subject.

List of Exclusion Criteria:

1. The subject has used topical or systemic therapies that might interfere with the evaluation of the study medication during the study.
2. The subject has a history of hypersensitivity to any of the ingredients in the study medication formulations.
3. The subject is unable to return for follow-up tests.
4. The subject has uncontrolled systemic disease, including known HIV positive patients.
5. The subject has a history of other skin conditions or significant illness that would interfere with evaluation of the study medication.
6. Any condition or situation which in the Investigator's opinion may put the subject at significant risk, could confound the study results, or could interfere significantly with the subject's participation in the study.
7. The subject has a history of invasive cancer within the past five years excluding non-melanoma skin cancer, Stage I cervical cancer, or CLL Stage 0.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ervin Epstein, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland; David R. Bickers, MD, Principal Investigator — Herbert Irving Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Children's Hospital and Research Center Oakland, Oakland, California
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York

REFERENCES:
- [Result] Tang JY, Chiou AS, Mackay-Wiggan JM, Aszterbaum M, Chanana AM, Lee W, Lindgren JA, Raphael MA, Thompson BJ, Bickers DR, Epstein EH Jr. Tazarotene: randomized, double-blind, vehicle-controlled, and open-label concurrent trials for basal cell carcinoma prevention and therapy in patients with basal cell nevus syndrome. Cancer Prev Res (Phila). 2014 Mar;7(3):292-9. doi: 10.1158/1940-6207.CAPR-13-0305. Epub 2014 Jan 17. PMID 24441673

RESULTS

PARTICIPANT FLOW:
Groups:
- Tazarotene Cream: This is a 36 month, multi-center, single arm, open label clinical study design
Period: Overall Study
Arm/Group | Tazarotene Cream
Started | 36
Completed 18 Months | 23
Completed | 13
Not Completed | 23

BASELINE CHARACTERISTICS:
Arm/Group | Tazarotene Cream
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: The primary endpoint used to evaluate tazarotene efficacy for BCC chemotherapy was the complete response (CR) rate, defined as the complete visible disappearance of a patient's "target" lesion during the the 18 months of tazarotene application and its failure to recur during the ensuing 18-months. We defined surgical removal of a target lesion as a treatment failure. The primary endpoint was assessed based on intention to treat analysis such that any subject who underwent the baseline evaluation and applied at least 1 dose of tazarotene was included in the analysis. Drop-outs were considered non-responders. A priori treatment success for tazarotene was defined as a CR rate of at least 50%, and treatment failure was defined as a CR rate of 25% or less.
Time Frame: 36 months
Population: N=2 participants excluded from analysis: N=1 due to revised BCNS diagnosis and N=1 because unable to confirm administration of at least one dose of tazarotene.
Measure: Count of Participants; unit: Participants
Arm/Group | Tazarotene Cream
Number analyzed (Participants) | 34
Participants | 2

2. Secondary Outcome: Time to Lesion Clearance
Time Frame: 36 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tazarotene Cream
Number analyzed (Participants) | 34
Participants | NA — The PI has left the institution and the only access to the data is from the publication. The access to this specific data cannot be confirmed and is not available to be reported.

3. Secondary Outcome: Time to Progression
Time Frame: 36 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tazarotene Cream
Number analyzed (Participants) | 34
Participants | NA — The PI has left the institution and the only access to the data is from the publication. The access to this specific data cannot be confirmed and is not available to be reported.

4. Secondary Outcome: Estimated Duration of Complete Response
Time Frame: 36 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tazarotene Cream
Number analyzed (Participants) | 34
Participants | NA — The PI has left the institution and the only access to the data is from the publication. The access to this specific data cannot be confirmed and is not available to be reported.

5. Secondary Outcome: Overall Response at Treated Lesions
Time Frame: 36 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tazarotene Cream
Number analyzed (Participants) | 34
Participants | NA — The PI has left the institution and the only access to the data is from the publication. The access to this specific data cannot be confirmed and is not available to be reported.

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | Tazarotene Cream
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 2/36
Other Adverse Events (participants affected / at risk) | 31/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tazarotene Cream (N=36)
prostate cancer diagnosis (Renal and urinary disorders) | 1
cellulitis and maxillary sinusitis (Ear and labyrinth disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tazarotene Cream (N=36)
irritation (Skin and subcutaneous tissue disorders) | 6
dryness (Skin and subcutaneous tissue disorders) | 6
inflammation (Skin and subcutaneous tissue disorders) | 1
itching (Skin and subcutaneous tissue disorders) | 3
peeling (Skin and subcutaneous tissue disorders) | 4
edema (Skin and subcutaneous tissue disorders) | 1
rash (Skin and subcutaneous tissue disorders) | 4
erythema (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes